CLINICAL TRIAL: NCT02692898
Title: Biomarker Analysis of Central Nervous System Tumors
Status: Terminated | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999916069; 16-C-N069
Record Dates: First submitted 2016-02-25; First posted 2016-02-26 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11-15

CONDITIONS: Central Nervous System Neoplasms; Primary Brain Neoplasms; Neoplasms, Brain; Cancer of the Brain; Brain Cancer
Keywords: Brain Tumor; Molecular Pathology; Clinical Data; Imaging Data
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- 1: Archived CNS neoplasm specimens, in which primary diagnostic studies are complete, and for which there is excess tissue for analysis in the form of unstained slides or paraffin blocks

SUMMARY:
Background:

The number of people who get tumors of the brain or central nervous system (CNS) is lower than other cancers. But these tumors cause a higher rate of serious effects and even death. Researchers want to test existing samples of tissue from these tumors to learn more about them. This may lead to better treatment.

Objective:

To study stored samples of CNS tumors to learn more about the tumors and explore new ways to diagnose them.

Eligibility:

The study will use tissue samples already collected at NIH from people with brain or CNS tumors.

Design:

The participants will have given their consent in a previous study.

Researchers will review the tissue samples and any data collected about them.

Researchers will do lab tests and scans on the samples.

All data will be kept secure.

DETAILED DESCRIPTION:
BACKGROUND

* Central Nervous System (CNS) and brain tumors are a heterogeneous group of neoplasms. They can be broadly categorized to tumors of neuroepithelial tissue, meninges, hematopoietic system, germ cells, and sella.
* The Central Brain Tumor Registry of the United States reports an overall average annual age-adjusted incidence rate for the years 2006-2010 for primary brain and CNS tumors as 21.03 per 100,000. This leads to an estimated mortality of over 13,000 deaths per year. Although this number is small compared to other more common cancers, due to the location of CNS (brain and spinal cord) tumors, they are responsible for disproportionately high morbidity and mortality among cancer patients.
* Although much progress has been made on overall understanding of CNS tumors, not much is known about mechanisms responsible for intratumoral heterogeneity, disease relapse, progression into higher grades, and in vivo invasive mechanisms. This may involve new mutations, selection of specific clones of cells by either therapeutic pressure or as part of natural tumor evolution leading to progression, microenvironmental cues or combinations.
* This study will review the molecular pathological alterations of archived human CNS tumor specimens at initial presentation and at subsequent relapse. We will request archived brain tumor tissue samples from the NCI CCR Laboratory of Pathology at multiple time points to determine the expression of cellular proteins and surrogate markers involved in growth, proliferation, differentiation, invasion, and survival of brain tumor cells. Such information will be pooled with imaging data (MRI, PET, etc.) to identify potential surrogate markers of disease resistance.
* This study has the potential to uncover key molecular events underlying disease progression and thereby contribute to the understanding of CNS tumor pathogenesis without active patient intervention.

OBJECTIVES

-To study archived specimens of CNS tumors from the NCI CCR Laboratory of Pathology to explore potential new biomarkers for diagnosis and to better understand CNS tumor pathogenesis.

ELIGIBILITY

* Diagnosis of CNS neoplasm.
* Eligible cases include those in which primary diagnostic studies are complete, and for which there is excess tissue for analysis in the form of unstained slides or paraffin blocks archived in the NCI CCR Laboratory of Pathology as well as imaging stored in the NIH medical records system.
* We also request permission to extend this analysis, as may be relevant in the future, to surplus materials to be accrued under existing NCI protocols, upon completion of all superseding diagnostic tests and medical/scientific studies.

DESIGN

* We anticipate obtaining approximately 500 archived specimens in the NCI CCR Laboratory of Pathology from patients with CNS neoplasms to analyze parameters in order to better understand the biology and pathogenesis of disease.
* To identify potential specimens, medical records of patients seen in the Neuro-Oncology and Neurosurgery Clinics will be reviewed. Additional medical records will be reviewed in order to identify archived specimens and to obtain ancillary information such as result of imaging studies.
* Existing biomarker data will be analyzed in conjunction with review of histological features and clinical data existing in laboratory and imaging data to arrive at improved criteria for diagnosis, and to recognize newly identified, as yet undescribed, disease entities. New biomarkers, as they may become available, will be utilized to improve on current diagnostic methods for disease definition.
* Tissue may be collected from pathology to be processed for specific research question at a future time point. Time of processing may be contingent on accumulating sufficient number of specimens.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:
* Diagnosis of CNS neoplasm.
* Eligible cases include those in which primary diagnostic studies are complete, and for which there is excess tissue for analysis in the form of unstained slides or paraffin blocks archived in the NCI CCR Laboratory of Pathology as well as imaging stored in the NIH medical records system. Cases will be drawn from specimens previously submitted to the NCI CCR Laboratory of Pathology in consultation or from surplus materials from existing protocols, upon completion of all superseding diagnostic tests and medical/scientific studies in cases where the patient is deceased or has previously consented to future use of samples on their original protocol consent. Inclusion of additional NIH cases will be limited to those instances in which the current informed consent encompasses the proposed analyses.

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-02-25; Primary Completion 2019-11-15 (Actual); Study Completion 2019-11-15 (Actual)

PRIMARY OUTCOMES:
Tumor profile of CNS Tumors | completion of study
  To study archived specimens of CNS tumors from the NCI CCR Laboratory of Pathology to explore potential new biomarkers for diagnosis and to better understand CNS tumor pathogenesis.

CONTACTS AND LOCATIONS:
Overall Officials: Terri S Armstrong, C.R.N.P., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute (NCI), 9000 Rockville Pike, Bethesda, Maryland, United States